CLINICAL TRIAL: NCT04241744
Title: Prospective, Randomized, Double-Blind, Trial of Oral Vancomycin Therapy Compared to Placebo As Primary Prevention for C. Difficile-associated Infection (CDI)
Brief Title: Prospective Trial of Oral Vancomycin Therapy vs. Placebo for Prevention of CDI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty enrolling patients
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Christopher Destache, Professor, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2000200-01
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: CDI
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- vancomycin oral solution (Active Comparator): vancomycin oral solution will be administered to consented patients >65 years of age receiving IV antimicrobial(s) for a bacterial infection twice daily while hospitalized.
  Interventions: Drug: Vancomycin 125 MG po BID
- placebo oral solution (Placebo Comparator): placebo oral solution will be administered to consented patients >65 years of age receiving IV antimicrobial(s) for a bacterial infection twice daily while hospitalized.
  Interventions: Drug: Vancomycin 125 MG po BID

INTERVENTIONS:
Drug: Vancomycin 125 MG po BID — prevention to develop CDI during hospitalization
  Other Names: placebo oral solution po BID

SUMMARY:
The purpose of this research study is to determine in patients receiving intravenous (IV) antibiotic(s), if giving oral vancomycin therapy will prevent C. difficile-associated infection (commonly called CDI). Oral vancomycin is an antibiotic that is commonly used to treat CDI. The investigators want to study if using this drug can prevent the development of CDI while you are in the hospital receiving IV antibiotics. The key risk factors for developing CDI are age and IV antibiotic therapy. CDI is an infection in your colon caused by an organism called Clostridium difficile (or C. diff for short) that causes diarrhea. Up to 12% of hospital-acquired infections have been reported to be CDI. It can lead to longer hospital stays and more costs associated with the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* 1. Older patients (> 65 years of age), hospitalized for > 48 hours and treated with parenteral antimicrobial therapy for > 48 hours at CHI Creighton University Medical Center-Bergan Mercy will be eligible for enrollment.

Exclusion Criteria:

1. Patients diagnosed with CDI within the first 72 hours of hospitalization and/or diagnosed with CDI within the past 3 months
2. Patients diagnosed with gastrointestinal infection other than CDI
3. Patients who have received a solid-organ transplant in the past 12 months
4. Females who are pregnant or immediately post-partum
5. Patients admitted to the hospital with an opportunistic infection secondary to HIV-1 and CD4 cell count of < 200 cell/mm3
6. Patients receiving cancer chemotherapy or immune modulator drugs (i.e. Checkpoint inhibitors; PD-1/PD-L1 inhibitors; biologic DMARDs) as examples
7. Patients being treated with ≥ 28 days of intravenous (IV) antimicrobials (complex S. aureus bacteremia, osteomyelitis, endocarditis)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
number of enrolled patients who develop CDI during hospitalization assessed ("up to 3 month") | during hospitalization through study completion, assessed up to 3 months
  number of enrolled patient with CDI receiving oral vancomycin compared to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University Medical Center - Bergan Mercy, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No